CLINICAL TRIAL: NCT04794738
Title: A Phase II/III, Randomized, Double-Blind, Placebo- and Active-controlled Study of SHR8554 Injection for the Treatment of Pain After Orthopedic Surgery
Brief Title: A Clinical Study of SHR8554 Injection for the Treatment of Pain After Orthopedic Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR8554-202
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Saline Solution; Morphine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A (Experimental)
  Interventions: Drug: SHR8554
- Treatment group B (Experimental)
  Interventions: Drug: SHR8554
- Treatment group C (Placebo Comparator)
  Interventions: Drug: Saline Solution
- Treatment group D (Active Comparator)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: SHR8554 — SHR8554 Injection; high dose
  Arms: Treatment group A
Drug: SHR8554 — SHR8554 Injection; low dose
  Arms: Treatment group B
Drug: Saline Solution — Saline Solution
  Arms: Treatment group C
Drug: Morphine — Morphine
  Arms: Treatment group D

SUMMARY:
The primary objective is to evaluate the analgesic efficacy of IV SHR8554 compared with placebo and morphine in patients with acute postoperative pain following orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Subjects requiring elective general anesthesia orthopedic surgery
3. Conform to the ASA Physical Status Classification

Exclusion Criteria:

1. Subjects with a history of difficult airway
2. Subjects with a history of reflux esophagitis
3. Subjects with a history of mental illness
4. Subjects with poor blood pressure control
5. Transcutaneous oxygen saturation (SpO2) <90%
6. Random blood glucose ≥11.1mmol/L
7. Subjects with abnormal liver function
8. allergies to opioids and other medications that may be used during the trial
9. Pregnant or nursing women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2021-04-18 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
the Sum of Pain Intensity Differences in Pain Score Over 48 Hours in the rest state | 48-hours
  Pain intensity will be evaluated using an 11-point (0-10) Numeric Pain Rating Scale (NPRS), with higher numbers indicating a higher pain intensity, administered over 48 hours. Time weighted average change from baseline is calculated using the following: time weighted sum of pain intensity differences (SPID) divided by a constant (48 hours) to yield values on the 0-10 NPRS.

SECONDARY OUTCOMES:
the Sum of Pain Intensity Differences in Pain Score Over 6、12、48 、12-24、24-48 Hours under static condition | 48-hours
the Sum of Pain Intensity Differences in Pain Score Over 6、12、24、48 、12-24、24-48 Hours under moving condition | 48-hours
Time of first use of remedial analgesic medication | 48-hours
Cumulative use of remedial analgesics from 0h to 48h | 48-hours
Participant ' satisfaction score for analgesia treatment | 48-hours
Investigator satisfaction score for analgesia treatment | 48-hours

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiaotong University School of Medicine,Renji Hospital, Shanghai, Shanghai Municipality, China